CLINICAL TRIAL: NCT06231069
Title: Effects of Mixed Exercise Training and a Novel Multi-Nutrient Supplement on Muscle Fitness in Young Adults
Brief Title: Mixed Exercise Training and Novel Multi-Nutrient Supplementation in Young Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19: Study halted prior to enrollment of first participant.
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 7405
Record Dates: First submitted 2019-07-12; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sarcopenia
Keywords: Muscle
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The present study is a randomized, double-blind, placebo-controlled 12-week mixed training and supplementation study (placebo vs. active supplement), with data collection occurring at several different time-points (pre, mid, and post) in young males and females (18-30 years of age).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following stratification (balanced by age, gender, dietary patterns, and PA levels), randomization into supplement vs. placebo groups will be done by an outside party. Thereafter, GCP (good clinical practice)-certified research coordinators will administer the supplements and collect the baseline/post data in a blinded fashion. These data will be locked and the code for randomization will not be broken until the study is completed. The integrity of the data and the quality of the data analyses will be verified by an outside source. Compliance to GCP will be checked regularly throughout the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-nutrient supplementation during training (Experimental)
  Interventions: Dietary Supplement: Multi-nutrient supplement; Other: Exercise
- Placebo during training (Placebo Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Dietary Supplement: Multi-nutrient supplement — 12 weeks of supplement intake of milk proteins, N-3 PUFAs, creatine, and vitamin D at levels previously shown to augment muscle protein synthesis in young individuals.
  Arms: Multi-nutrient supplementation during training
Other: Exercise — 12 weeks of short-duration mixed endurance and resistance exercise.

SUMMARY:
This study aims to elucidate the effects of 12 weeks of novel multi-nutrient supplementation combined with mixed aerobic/resistance exercise training on skeletal muscle function in young adults.

It is hypothesized that multi-nutrient supplementation and mixed aerobic/resistance exercise training (AET/RET) will have interactive effects on muscle fitness.

DETAILED DESCRIPTION:
Sedentarism is highly prevalent, world-wide, and predisposes for chronic disease and premature death. Conversely, regular physical activity (PA) protects against cardiovascular disease (CVD), deterioration of the musculoskeletal system, cancer, obesity, type 2 diabetes, depression, anxiety, and neurodegeneration. Similar to most adults in the world, the majority of Canadians are not meeting the minimal PA guidelines, with total health care cost attributed to physical inactivity estimated to be $6.8 billion. Therefore, it is imperative to develop strategies to increase PA rates across the general population (young to old) to alleviate the global burden of chronic disease. These strategies may include large-scale, societal interventions that incentivize daily PA/sports participation (mainly access and affordability), educational efforts, and continued support of exercise science research. Specifically, research on exercise modes that are time-saving but equally (or more) effective as traditional training modes is warranted. More studies are also needed on nutritional supplementation (safety and efficacy), particularly in conjunction with various exercise modes for optimization of health and performance.

In this randomized, double-blind, placebo-controlled clinical trial, the aim is to elucidate the effects of 12 weeks of novel multi-nutrient supplementation combined with mixed aerobic/resistance exercise training on skeletal muscle function in young adults. Following recruitment, participants will be stratified and randomized into one of four groups:

1. Healthy, recreationally active young males, placebo, n = 15
2. Healthy, recreationally active young males, multi-nutrient supplement, n = 15
3. Healthy, recreationally active young females, placebo, n = 15
4. Healthy, recreationally active young females, multi-nutrient supplement, n = 15

Thereafter, subjects will undergo 12 weeks of a mixed AET and RET, three days per week, approximately 1 hour per training session. The AET will consist of cycle ergometry for 20 min at 75% HRmax, corresponding to ~65% VO2max (Monark cardio care 827E). As the aerobic fitness of the subjects are progressively enhanced, the cadence RPM and/or resistance of the bike will be increased to elicit 65% VO2max. This work rate, corresponding to ~75% HRmax, will be monitored by the subjects wearing a heart rate monitor around their chests (Polar). Immediately following the AET, the subjects will perform a lower body resistance exercise program consisting of four traditional resistance exercises starting at 65% of 1-RM (Cybex Eagle). Specifically, the RET program will consist of leg press, seated calf extension, knee extension, and hamstring curls, to be performed at 65% 1-RM for 4 x 15 repetitions initially, and thereafter progressively increased throughout the 12-week intervention period to 85% 1-RM for 4 x 8 repetitions. Resistance will be increased with ~2-10% in load when the individual can perform the current workload for one or two repetitions over the desired number on two consecutive training sessions. Prior to beginning the research coordinator will meet with participants and teach them how to properly perform exercises (familiarization session).

Concurrently, participants will be asked to consume 7 servings of a multi-nutrient supplement per week with 200 mL water. The supplement consists of mixed milk proteins, creatine, N-3 PUFAs, and vitamin D at levels previously shown to stimulate muscle protein synthesis. On training days, the compound will be consumed immediately after the training session under the supervision of a study coordinator. On the remaining four days, subjects will consume 1 serving prior to breakfast, which is regarded as the least protein-rich meal of the day. In order to monitor 'at-home' compliance, the subjects will be instructed to record their daily intake in a supplement log.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* non-diabetic
* apparently healthy
* minimally recreationally active
* males and females aged 18-30 years

Exclusion Criteria:

* pregnancy
* breast feeding
* smoking
* obesity
* diabetes mellitus
* cardiovascular disease (recent myocardial infarction (≤ 6 months)
* hypertension requiring more than 2 medications
* congestive heart failure requiring more than one medication,
* renal disease (creatinine > 130),
* previous stroke with residual hemiparesis,
* active musculoskeletal injuries and/or severe osteoarthritis,
* significant weight loss in the 3-month period prior to the study,
* vegan diet,
* dairy protein allergy,
* muscular dystrophy,
* severe peripheral neuropathy,
* severe osteoporosis,
* use of medications known to affect protein metabolism (i.e. corticosteroids),
* inability to consent,
* chronic obstructive pulmonary disease (FVC or FEV1 < 70% of age predicted mean value),
* asthma requiring more than two medications.
* Subjects on supplements will be considered on a case-by-case basis, but they will be asked to refrain from intake for at least 2 weeks prior to partaking in this study.
* While adverse events are not anticipated, participants will be asked to disclose if they are using supplements that may have negative/interactive effects with our study products. Each participant's list of medications will also be checked for potential interactive side-effects with our supplements; however, the individual doses have specifically been chosen to be at the low end to minimize the likelihood of such interactions.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2030-01-20 (Estimated); Primary Completion 2030-04-20 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Percent change in DXA-obtained muscle mass | 12 weeks
  Pre to post change in DXA-obtained muscle mass (%)
Percent change in DXA-obtained fat mass | 12 weeks
  Pre to post change in DXA-obtained fat mass (%)
Percent change in DXA-obtained muscle mass to fat mass ratio | 12 weeks
  Pre to post change in DXA-obtained muscle mass to fat mass ratio (%)
Percent change in bodyweight | 12 weeks
  Pre to post change in bodyweight (%)
Percent change in body mass index | 12 weeks
  Pre to post change in body mass index (%)
Percent change in waist to hip ratio | 12 weeks
  Pre to post change in waist to hip ratio (%)

SECONDARY OUTCOMES:
Percent change in slow muscle fiber areas | 12 weeks
  Pre to post change in slow muscle fiber areas (%)
Percent change in fast muscle fiber areas of quadriceps | 12 weeks
  Pre to post change in fast muscle fiber areas of quadriceps (%)
Percent change in quadriceps circumference | 12 weeks
  Pre to post change in quadriceps circumference (%)
Percent change in essential amino acid blood levels | 12 weeks
  Pre to post change in venous essential amino acid blood levels (%)
Percent change in inflammatory cytokine blood levels (interluekins) | 12 weeks
  Pre to post change in venous inflammatory cytokine blood levels (interleukins) (%)
Percent change in maximal leg extension strength | 12 weeks
  Pre to post change in leg extension (%)
Percent change in maximal leg press strength | 12 weeks
  Pre to post change in maximal leg press strength (%)
Percent change in number of repetitions at 60% maximum in leg press | 12 weeks
  Pre to post change in number of repetitions at 60% maximum in leg press (%)
Percent change in maximal aerobic capacity | 12 weeks
  Pre to post change in maximal aerobic capacity (%)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Tarnopolsky, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No